CLINICAL TRIAL: NCT07215078
Title: A PHASE 1, OPEN-LABEL, TWO-PERIOD, CROSS-OVER STUDY TO EVALUATE DOSE PROPORTIONALITY OF ATIRMOCICLIB (PF-07220060) PHARMACOKINETICS WHEN ADMINISTERED UNDER FED CONDITIONS TO HEALTHY PARTICIPANTS
Brief Title: Study About Whether Atirmociclib/PF-07220060 Proportionally Increases Exposure as Dose Increases in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C4391030
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer
Keywords: Dose proportionality on the pharmacokinetics; Dose proportionality on the safety and tolerability; Atirmociclib (PF-07220060)

STUDY DESIGN:
Intervention Model Description: Phase 1, open-label, randomized, two-period, cross-over study to evaluate the dose proportionality on the pharmacokinetics, safety, and tolerability
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1 (Experimental): In Period 1 Day 1, participants from Sequence AB and BA will receive Dose A and Dose B atirmociclib higher drug load IR MST tablet, respectively.
  In Period 2 Day 1, the participants from two sequences in the same cohort will shuffle the treatment.
  Interventions: Drug: atirmociclib (PF-07220060)
- Cohort 2 (Experimental): In Period 1 Day 1, participants from Sequence AC and CA will receive Dose A and Dose C atirmociclib higher drug load IR MST tablet, respectively.
  In Period 2 Day 1, the participants from two sequences in the same cohort will shuffle the treatment.
  Interventions: Drug: atirmociclib (PF-07220060)
- Cohort 3 (Experimental): In Period 1 Day 1, participants from Sequence BC and CB will receive Dose B and Dose C atirmociclib higher drug load IR MST tablets, respectively.
  In Period 2 Day 1, the participants from two sequences in the same cohort will shuffle the treatment.
  Interventions: Drug: atirmociclib (PF-07220060)
- Cohort 4 (Experimental): In Period 1 Day 1, participants from Sequence AD and DA will receive Dose A and Dose D atirmociclib higher drug load IR MST tablet, respectively.
  In Period 2 Day 1, the participants from two sequences in the same cohort will shuffle the treatment.
  Interventions: Drug: atirmociclib (PF-07220060)
- Cohort 5 (Experimental): In Period 1 Day 1, participants from Sequence BD and DB will receive Dose B and Dose D atirmociclib higher drug load IR MST tablets, respectively.
  In Period 2 Day 1, the participants from two sequences in the same cohort will shuffle the treatment.
  Interventions: Drug: atirmociclib (PF-07220060)
- Cohort 6 (Experimental): In Period 1 Day 1, participants from Sequence CD and DC will receive Dose C and Dose D atirmociclib higher drug load IR MST tablets, respectively.
  In Period 2 Day 1, the participants from two sequences in the same cohort will shuffle the treatment.
  Interventions: Drug: atirmociclib (PF-07220060)

INTERVENTIONS:
Drug: atirmociclib (PF-07220060) — Open-label, two-period, cross-over study to evaluate dose proportionality of atirmociclib (PF-07220060) pharmacokinetics when administered under fed condition to healthy participants

SUMMARY:
The purpose of this clinical trial is to learn about the dose proportionality on the PK of the study medicine (called atirmociclib) when administered in the various doses range under the fed condition in healthy participants.

This study is seeking participants who are:

1. male and female aged 18 to 65 years are healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests
2. with BMI of 17.5-30.5 kg/m2; and a total body weight >50 kgs (110 lbs.).

All participants (72 total) in this study will receive atirmociclib at Dose (A), Dose (B), Dose (C), and Dose (D) oral dose in 1 of the 12 treatment sequences among 6 cohorts under fed conditions.

Atirmociclib will be given by mouth at the study research unit once single dose about 30 minutes after a moderate fat standard calorie meal.

Dose proportionality will be evaluated on the pharmacokinetics (PK), safety and tolerability of atirmociclib at Doses (A), (B), (C), and (D) oral dose under the fed condition.

Including the 28 days of screening window and the 35 days safety follow-up period, the total study duration for each participant can be up to 71 days, containing 2 periods (6 days for each period), minimum 7-day interval between two periods, and follow-up period 28 to 35 days from administration of the final dose of study intervention. During this time, they will undergo safety laboratory and serial blood PK samplings up to 120 hours after administration of atirmociclib to determine plasma concentrations of atirmociclib. Participants will be discharged from the research unit on Period 2 Day 6 following completion of all assessments.

ELIGIBILITY:
Inclusion:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
* Body mass Index (BMI) of 17.5-30.5 kg/m2; and a total body weight >50 kg (110 lb.).

Exclusion:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* Concomitant use of any medications or substances that are strong inducers or inhibitors of CYP3A4 or UGT2B7 are prohibited within 5 half-lives plus 14 days (up to 28 days) prior to first dose of atirmociclib.
* Previous exposure to atirmociclib or participation in studies requiring atirmociclib administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | 1 hour prior to atirmociclib dosing, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose
  Dose-normalized plasma AUCinf and Cmax of atirmociclib for each cohort (AUClast if AUCinf cannot be estimated)
Maximum Observed Plasma Concentration (Cmax) | 1 hour prior to atirmociclib dosing, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) by Seriousness and Relationship to Treatment | Period 1: Days 1-6; minimum 7-day interval between two doses; Period 2: Day 1-35
Number of Participants With Laboratory Abnormalities | Period 1: Days 1-6; minimum 7-day interval between two doses; Period 2: Day 1-35
Number of Participants With Abnormalities in Physical Examination | Period 1: Days 1-6; minimum 7-day interval between two doses; Period 2: Day 1-35
Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Findings | Period 1: Days 1-6; minimum 7-day interval between two doses; Period 2: Day 1-35
Number of Participants With Concomitant Medications | Period 1: Days 1-6; minimum 7-day interval between two doses; Period 2: Day 1-35

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4391030